CLINICAL TRIAL: NCT03974399
Title: Longitudinal Assessment of BDNF Levels in Healthy Subjects Taking Bacopa Monnieri
Brief Title: BDNF Levels After Bacopa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roskamp Institute Inc. (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RI-Bacopa-001
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2019-06

CONDITIONS: Memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study enrollment (Other): all participants will take dietary supplement, Bacopa Monnieri, daily for 3 months
  Interventions: Dietary Supplement: Bacopa Monnieri

INTERVENTIONS:
Dietary Supplement: Bacopa Monnieri — subjects will take Bacopa Monnieri daily for 3 months

SUMMARY:
Brain-derived neurotrophic factor (BDNF) is a well-known neurotrophic factor important for learning, memory, and synaptogenesis. Healthy activities such as exercise are believed to raise BDNF, while stress is associated with lower BDNF. What is not well understood is if there are certain supplements that may raise BDNF over time. Bacopa monnieri is well characterized nutraceutical. Animal and pre-clinical data support multiple beneficial mechanisms, including raising BDNF and increasing synaptogenesis. Additionally, small studies have shown Bacopa enhances cognition and improves mood. We would like to investigate if BDNF level changes in people after starting Bacopa.

DETAILED DESCRIPTION:
This is a single site two-visit, 12-week, open label, trial to evaluate the safety, tolerability, and potential effects of Bacopa on BDNF, MoCA and GDS. Potentially eligible subjects will be invited to screening (Visit 1) at the study site. Subjects will sign an informed consent followed by collection of medical history and history of current medications, have their height, weight, vital signs (blood pressure, pulse, and temperature) measured, complete study assessments (MoCA , BDS and LEC) Routine clinical laboratory tests (hematology and chemistry) will be performed. Blood samples will be taken for analysis of BDNF and genetics (APOE, BDNF).

Subjects will be instructed to orally self-administer the provided supplement (Bacopa) preferably with food with no dietary restrictions once a day in the morning.

Subjects will be contacted by phone at 1 week (+/- 3 days) to be reminded to go to two pills per day, 1 month (+/-1 week) to check on compliance or any AE's and 2 months (+/- 1 week) to report any Adverse events for review by the Principal Investigator.

Subjects will return to the study site for Visit 2 at the end of 12 weeks (+/- 1 week). Study staff will question subjects about any changes in the subject's health since the first visit. They will be asked about their exercise activity and if there have been any changes to their LEC-5. Subjects will have their weight and vital signs measured. Routine clinical laboratory tests (hematology and chemistry) will be performed, and blood samples will be saved for analysis of Bacopa and other biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of any ethnicity, at 60 to 78 on day of screening.
2. Have a score of 25 or above on MoCA (Montreal Cognitive assessment).
3. Have a score of 9 or below on GDS (Geriatric Depression Scale)
4. Provide written informed consent.
5. Be able and willing to follow instructions, participate in study assessments, and be present for the required study visits.
6. Otherwise stable medical history and general health up to the discrepancy of the PI.

Exclusion Criteria:

1. Have contraindications, allergy, or sensitivity to the study product or their components.
2. Have any significant illness or condition that could, in the Investigator's or sub-Investigator's opinion, be expected to interfere with the study parameters or study conduct or put the subject at significant risk. These may include but are not limited to: untreated chronic hypertension; receiving chemotherapy; depression requiring medical intervention on a daily basis; myocardial infarction within six months of screening; renal failure; and/or hepatic failure.
3. Have a current unstable medical condition (e.g., symptomatic uncontrolled diabetes mellitus), or a condition that might affect their ability to participate (e.g., cancer requiring frequent medical visits for chemotherapy).
4. Have values on standard clinical laboratory assessments that are deemed medically significant (show evidence of untreated significant medical illness or pose a risk of significant intercurrent illness during the study in the opinion of the investigator).
5. Currently taking any medication classified by the FDA as an anti-depressant or have discontinued one of these types of medications within 30 days of screening.
6. Currently abusing drugs or alcohol, and/or have a history of drug or alcohol dependence within six months of entering this study.

Ages: 60 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Brain Derived neurotrophic factor (BDNF) | 3 months
  a. Change in BDNF levels
Changes in Brain Derived Neurotropic factor (BDNF) signaling pathway | 3 months
  Change in BDNF signaling pathway

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment | 3 months
  Changes in Montreal Cognitive Assessment (MoCA). Score range 0-30.
Change in Geriatric Depression Scale | 3 months
  Change in Geriatric Depression Scale (GDS). Score range 0-15.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Keegan, M.D., Principal Investigator — The Roskamp Institute Inc
Locations (1):
- The Roskamp Institute, Inc., Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No